CLINICAL TRIAL: NCT00474942
Title: Apparent Mineralocorticoid Excess Syndrome Natural History Clinical Protocol
Brief Title: Natural History of Apparent Mineralocorticoid Excess Syndrome
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); Rare Diseases Clinical Research Network (Network); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 04-0474; U54HD064382 (NIH); RDCRN 5601 (Other: Office of Rare Diseases (ORD))
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Apparent Mineralocorticoid Excess Syndrome
Keywords: Hypertension; Metabolic Alkalosis; Hypokalemia
MeSH Terms: conditions — Mineralocorticoid Excess Syndrome, Apparent; Hypertension; Hypokalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Apparent mineralocorticoid excess (AME) is a rare inherited disease that can cause severe high blood pressure and low blood potassium in children and adults. It is caused by abnormal hormone metabolism and can be fatal. This study will focus on the genetic basis, natural history, disease progression, and survival of people with AME.

DETAILED DESCRIPTION:
AME is a rare genetic disorder that is caused by a mutated HSD11B2 gene, which encodes the metabolic enzyme 11BHSD2. The altered gene interferes with the ability of 11BHSD2 to inactivate the hormone cortisol. Above-normal cortisol activity then leads to a rise in blood pressure and a reduction of potassium in the blood. It also leads to low levels of the enzyme renin and the hormone aldosterone, both of which are involved in the regulation of long-term blood pressure. Long-term high blood pressure and metabolic defects start at an early age in children with severe AME. In others, AME may start later in life and cause less serious side effects. Symptoms can include poor growth in childhood, delayed puberty, muscle weakness, heart rate irregularity, frequent urination, and thirst. If left untreated, AME can cause serious damage to the eyes, kidneys, heart, and other organs.

Current treatment with the synthetic steroid spironolactone usually improves symptoms; however, despite treatment, some individuals with AME still experience disease progression and even death within years of being diagnosed with AME. Understanding more about AME, how it progresses, and how it affects people differently may help to improve treatment options. The purpose of this study is to examine the genetic basis, natural history, disease progression, and outcome of children and adults with AME. The study will also examine the family members of study participants with AME for any genetic abnormalities and possible mild forms of AME.

This study will last 2 to 7 years. Participants and their family members will attend yearly study visits that will include interviews about medical history, symptoms, and hospital stays; a physical exam; blood pressure testing; and blood and urine collection. Interim reviews of medical records will occur as necessary. Children will undergo an x-ray of the left hand. During the initial study visit, participants will be asked questions about family members and birth size.

ELIGIBILITY:
Inclusion Criteria for Participants with AME:

* High blood pressure characterized by low plasma renin and serum aldosterone levels
* Elevated urinary cortisol/cortisone metabolite ratio ([THF + 5aTHF]/THE)
* Molecular genetic diagnosis of AME with two mutations of the HSD11B2 gene

Inclusion Criteria for Family Members without Genetic Diagnosis of AME:

* Carrier of the HSD11B2 mutation that the AME participant has

Exclusion Criteria for All Participants:

* Any other illness or condition that might interfere with study participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with apparent mineralocorticoid excess plus their family members
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2007-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria I. New, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (2):
  - Mount Sinai School of Medicine, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
- University of Sao Paulo, São Paulo, Brazil
- University of Lyon, Lyon, France

REFERENCES:
- [Background] New MI, Geller DS, Fallo F, Wilson RC. Monogenic low renin hypertension. Trends Endocrinol Metab. 2005 Apr;16(3):92-7. doi: 10.1016/j.tem.2005.02.011. PMID 15808805
- [Background] Palermo M, Quinkler M, Stewart PM. Apparent mineralocorticoid excess syndrome: an overview. Arq Bras Endocrinol Metabol. 2004 Oct;48(5):687-96. doi: 10.1590/s0004-27302004000500015. Epub 2005 Mar 7. PMID 15761540
- [Background] Quinkler M, Bappal B, Draper N, Atterbury AJ, Lavery GG, Walker EA, DeSilva V, Taylor NF, Hala S, Rajendra N, Stewart PM. Molecular basis for the apparent mineralocorticoid excess syndrome in the Oman population. Mol Cell Endocrinol. 2004 Mar 31;217(1-2):143-9. doi: 10.1016/j.mce.2003.10.019. PMID 15134813